CLINICAL TRIAL: NCT02140736
Title: Role of biOsimilaRs in Therapeutic Management of Anemia Following Chemotherapy in HEmatology and Oncology; A Prospective, Observational, Non-interventional Study
Brief Title: Epoetin Alfa Biosimilar in the Management of Chemotherapy-Induced Symptomatic Anemia in Haematology and Oncology
Acronym: ORHEO
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 1_09.04.2009; 09.214 (Other: CCTIRS)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2015-07

CONDITIONS: Chemotherapy-induced Symptomatic Anemia; Solid Tumors; Malignant Hemopathies; Lymphomas; Myelomas
Keywords: Chemotherapy-induced anemia; Epoetin biosimilar
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chemo-induced symptomatic anemia
  Interventions: Drug: Epoetin biosimilar

INTERVENTIONS:
Drug: Epoetin biosimilar

SUMMARY:
The main aim of this study is to observe correction of the hemoglobin level in the patients under chemotherapy, treated with epoetin alfa biosimilar and presenting with a solid tumor or a lymphoma or a myeloma.

DETAILED DESCRIPTION:
This is a non-interventional, descriptive, national, multi-site, longitudinal and prospective observational study with adults patients who are suffering from cancer or malignant blood disease and whose chemotherapy treatment has induced symptomatic anemia and being treated with biosimilar of epoetin to correct haemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 years of age
* Patients presenting with anemia following chemotherapy
* Patients suffer from solid tumours, malignant hemopathies, lymphomas or myelomas and presenting with anemia following chemotherapy

  -- The patients may be included regardless of their chemotherapy cycle (from the first cycle until the last cycle)
* Patients eligible for epoetin alfa biosimilar treatment

Exclusion Criteria:

* Patients are not receiving chemotherapy
* Patients already included in an epoetin zeta trial
* Patients presenting with a contraindication to epoetin zeta
* Patients presenting with hypersensitivity to the active principle or any of the excipients
* Patient with erythroblastopenia or acquired pure red cell aplasia (APRCA)
* Patient with uncontrollable arterial hypertension
* Patients who cannot receive adequate prophylaxis by antithrombotic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffer from solid tumours, malignant lymphomas or multiple myeloma and have developed symptomatic anaemia due to their chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 2333 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Change and corrected Hemoglobin levels | 6 months
  Participants who have hemoglobin values between 11 and 12 g/dl after 6 months of treatment.

SECONDARY OUTCOMES:
Observe evolution of the biological indicators | 6 months
  Observe evolution of the biological indicators: hemoglobin, hematocrit, reticulocytes, serum iron, ferritin, transferrin saturation
Study the profiles of treated patients | 6 months
Assess the reasons for the prescriber's treatment regimens | 6 months
Assess the correlations between the prescribing oncologists' treatment regimens and the patient characteristics | 6 months
Observation of the safety profiles of the Product (Epoetin Alfa) | 6 months

CONTACTS AND LOCATIONS:
Locations (119):
- France (119):
  - Agen
  - Aix-en-Provence
  - Ajaccio
  - Albi
  - Amboise
  - Amilly
  - Annecy
  - Antibes
  - Armentières
  - Arras
  - Aulnay-sous-Bois
  - Avignon
  - Bayonne
  - Beauvais
  - Besançon
  - Beuvry
  - Béthune
  - Béziers
  - Blois
  - Bois-Guillaume
  - Bordeaux
  - Boulogne-sur-Mer
  - Brest
  - Bron
  - Caen
  - Cannes
  - Carcassonne
  - Castelnau-le-Lez
  - Challes-les-Eaux
  - Chalon/saonne
  - Chambéry
  - Cherbourg-octeville
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Créteil
  - Croix
  - Désertines
  - Dijon
  - Draguignan
  - Dunkirk
  - Évreux
  - Feurs
  - Foix
  - Freyming-Merlebach
  - Fréjus
  - Fryming Merle BACH
  - Gap
  - Grasse
  - Haguenau
  - Hyères
  - La Roche-sur-Yon
  - La Rochelle
  - La Seyne-sur-Mer
  - La Tronche
  - Le Blanc-Mesnil
  - Le Mans
  - Lille
  - Limoges
  - Lyon
  - Mareuil LES MAUX
  - Marseille
  - Mâcon
  - Meaux
  - Metz
  - Monaco
  - Mont-de-Marsan
  - Montargis
  - Montauban
  - Montbéliard
  - Montfermeil
  - Montpellier
  - Morlaix
  - Moulins
  - Mulhouse
  - Nancy
  - Nantes
  - Nantes Saint Herblain
  - Narbonne
  - Nice
  - Niort
  - Nîmes
  - Nogent/Marne
  - Orléans
  - Paris
  - Perpignan
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Pontoise
  - Pringy
  - Reims
  - Rennes
  - Rouen
  - Saint-Cloud
  - Saint-Gaudens
  - Saint-Germain-en-Laye
  - Saint-Herblain
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Sainte-Feyre
  - Sélestat
  - Strasbourg
  - Talence
  - Tarbes
  - Thionville
  - Thonon-les-Bains
  - Toulon
  - Toulouse
  - Tours
  - Tremblay-en-France
  - Troyes
  - Valence
  - Vandœuvre-lès-Nancy
  - Versailles
  - Vénissieux
  - Vichy
  - Villefranche/saone
  - Villeneuve-sur-Lot

REFERENCES:
- [Derived] Michallet M, Luporsi E, Soubeyran P, Amar NA, Boulanger V, Carreiro M, Dourthe LM, Labourey JL, Lepille D, Maloisel F, Mouysset JL, Nahon S, Narciso B, Nouyrigat P, Radji R, Sakek N, Albrand H; ORHEO study group. BiOsimilaRs in the management of anaemia secondary to chemotherapy in HaEmatology and Oncology: results of the ORHEO observational study. BMC Cancer. 2014 Jul 10;14:503. doi: 10.1186/1471-2407-14-503. PMID 25011615